CLINICAL TRIAL: NCT00203242
Title: An Open-label Pilot Study to Collect/Evaluate Data on the Use of Consecutive Daily Intravenous Doses of Depacon in Combination With Daily Dose of Depakote ER During a Cluster Headache Cycle.
Brief Title: An Open Label Study Using Consecutive Intravenous Depacon With Oral Depakote ER for the Treatment of Cluster Headaches.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Stephen D. Silberstein, M.D.- Principal Investigator, Thomas Jefferson University/Jefferson Headache Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDS/DEP/01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Valproic Acid

ARMS (1):
- Depacon IV and Depakote ER (Experimental): Subjects will be treated in this single arm study with 2 consecutive days of IV Depacon followed by oral Depakote ER for a total of 1000 mg of Depacon and 1000 mg of Depakote ER each day.
  Interventions: Drug: Depacon IV and Depakote ER

INTERVENTIONS:
Drug: Depacon IV and Depakote ER

SUMMARY:
The purpose of this study is to collect and evaluate information on the use of Depakote Extended Release (ER) and Depacon Intravenous (IV) in patients with cluster headaches. Patients who are currently in a cluster cycle will be treated with 2 consecutive days of IV Depacon followed by oral Depakote ER. Patients will receive a total of 1,000mg of Depacon and 1,000mg of Depakote ER each day. Patients may have a 3rd day of IV Depacon followed by oral Depakote ER if the primary investigator believes it to be beneficial. The patient is then sent home on oral Depakote ER. The dose of Depakote ER can range from 500mg to 2,000mg this dose is to be determined by the primary investigator. The patient will continue the oral Depakote ER until the end of their cluster cycle or for a maximum of 6 weeks, which ever comes first.

DETAILED DESCRIPTION:
This study will consist of four visits (3 visits if the screening visit and first treatment visit are on the same day).

Screening Visit:

The screening visit can be performed either before an active cluster period or once the cluster period has already started. If the subject agrees to participate, the study doctor will determine if they are eligible for this study. The subject will be asked about their headache history, and medical history including all medications they are currently taking. A brief physical examination and neurologic examination will be performed and vital signs (pulse and blood pressure) will be measured. If the subject is a woman who is capable of bearing children, they will be asked to provide a urine sample for a routine pregnancy test. A blood sample (approximately 2 teaspoons) will also be obtained. Blood samples will be taken for a liver function test (LFT), complete blood count (CBC) with differential, chemistry profile, prothrombin time (PT) and partial thromboplastin time (PTT).If the screening visit is the same day as the first treatment visit, this blood work will be sent for immediate analysis. The results must be reviewed and approved by the study physician prior to the subject being administered study medication.

Treatment Visit One:

If the subject does not undergo treatment at the screening visit because they are not in an active cluster period, the subject will be asked to contact the site once their next cluster period begins. Subjects will be scheduled to come for their first treatment visit as soon as possible.

If the screening visit is not the same day as the first treatment visit, the study physician and or delegated research staff will re-explain the informed consent, ask the subject to re-read the informed consent and verbally re-confirm their agreement to participate in this trial.

The research staff will then determine whether the subject continues to qualify for the research trial. They will ask the subject about any changes in their medications since their last visit and/or any changes in their medical conditions since their last visit. Vital signs will be measured and if the subject is a woman of childbearing potential a urine sample will be obtained for routine pregnancy testing. A brief physical examination and neurologic examination will be performed by the study physician. The subject will be given a diary to take home with instructions on how to complete it. The subject will be scheduled to return to the study office the next day.

Once all of the above procedures have been completed, the research staff will then ask the subject to lie down in an exam room. They research nurse or study physician will then administer one of the study medications (Depacon) through an IV placed in their arm. Subjects will receive 1000mg of Depacon IV. This medication will be infused (administered) over a five minute period. The subjects' vital signs will be measured at 3 minutes, 5 minutes and 15 minutes after the medication has been completely administered.

The subject will remain in the study office for one hour for observation. Subjects will be closely monitored and repeatedly queried for the development of adverse events. Appropriate intervention and follow-up will be applied as deemed necessary by the investigator.

Prior to leaving the office, the research nurse or study physician will give the subject an oral dose of the second study medication, 1000mg of Depakote ER.

Treatment Visit Two:

The subject will return to the study office the next day for their second treatment visit. The study staff will review the subject's diary and record their vital signs. The subject's take home diary will be re-dispensed. The subject will then undergo the same infusion procedure as in their first treatment visit. Subjects will again receive a total of 1000mg of Depacon IV. Subjects will be closely monitored and repeatedly queried for the development of adverse events. Appropriate intervention and follow-up will be applied as deemed necessary by the investigator.

Prior to leaving the office, the research nurse or study physician will give the subject an oral dose of the second study medication, 1000mg of Depakote ER.

The subject may or may not be asked to return the next day for a third treatment day depending on the study physicians' review of their response to study treatment. If it is determined that the subject does not need to return for a third treatment day, a blood sample will be obtained from a vein in their arm. The subject will also be given a take home supply of the oral study drug Depakote ER with instructions. The subject will be scheduled to return to the study office in 6 weeks OR when their current cluster cycle ends, whichever comes first.

The research staff will contact the subject bi-weekly to see how they are doing and to confirm that they are taking your study drug appropriately. The research staff will also ask the subject if they have had any unwanted experiences since their last contact with the site. The subject will be instructed to call the study site should they have any questions or have any unwanted experiences.

Treatment Visit Three:

If the study physician determines that the subject should return for a third treatment day, the subject will return to the study office the day after their second treatment visit. The same infusion procedures will be performed. The study staff will review the subject's diary and record their vital signs. A blood sample (2 teaspoons) will be obtained from a vein in their arm. Prior to leaving the office, the research nurse or study physician will give the subject an oral dose of the second study medication, Depakote ER.

The subject will be given a take home supply of the oral study drug Depakote ER with instructions. Subjects will be instructed to take 2000mg of Depakote ER once a day. The subject will be scheduled to return to the study office in 6 weeks OR when their current cluster cycle ends, whichever comes first. The research staff will contact the subject bi-weekly to see how they are doing and to confirm that they are taking your study drug appropriately. The research staff will also ask whether or not the subject had any unusual symptoms, or out of the ordinary experiences since their last contact with the site. The subject will be instructed to call the study site should they have any questions or have any unwanted experiences.

Final Visit:

The final visit to the study office will occur either 6 weeks after the subjects last treatment visit OR when the subjects current cluster cycle ends, whichever comes first. At this visit, the study staff will collect and review the subject's diary as well as any unused study medication. The subject will be asked about any changes in medications and/ or medical conditions since their last contact with the site. The subject will also be asked about any unusual symptoms, or out of the ordinary experiences since their last contact with the site. The subject will be asked to report how they felt they responded to the study medication. The subject's vital signs will be measured and a blood sample (2 teaspoons) will be obtained from a vein in their arm.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 65 with a diagnosis of cluster headache (episodic or chronic) as defined by the International Headache Society criteria
* Subject is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female of child-bearing potential
* Subject has negative urine pregnancy test prior to study entry (Screening and Infusion Day 1), if female of child-bearing potential
* Subject is able to understand and comply with all study requirements
* Subject provides written informed consent prior to any screening procedures being conducted

Exclusion Criteria:

* Women who are pregnant or lactating
* Subjects who have a lifetime history of less than 2 cluster periods
* Subjects who have a typical cluster period of less than 6 weeks duration, or are currently in a cluster period that is expected to last less than 6 weeks from Infusion Day 1
* Subjects who have or have a history of hepatic conditions (such as hepatitis, liver failure or liver function tests (LFT's) greater than three times normal)
* Subjects who, in the investigators opinion, have a history or have evidence of a medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial
* Subjects who require a change in medication or existing regimen of medication in the 4 weeks prior to Infusion Day 1 and for the duration of the trial
* Subjects who require a change in medication or existing regimen of medication for the prophylaxis of cluster in the 4 weeks prior to Infusion Day 1 and for the duration of the trial
* Subjects who have used the following medications/ treatments from four weeks prior to Infusion Day 1: corticosteroids and nerve blocks.
* Subjects who are allergic to or have shown hypersensitivity to valproate or valproic acid
* Subjects with a history of significant drug or alcohol abuse within the past year
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit
* Subjects who have failed previous trials of Depakote or Depacon for the treatment of cluster headache

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-07; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Silberstein, MD, Principal Investigator — Thomas Jefferson University, Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Depacon IV and Depakote: Subjects will be treated with 2 consecutive days of IV Depacon (1000 mg/day) followed by oral Depakote ER (1000 mg/day). Subject continues oral Depakote ER until end of cluster cycle or for a maximum of 6 weeks, which ever comes first.
Period: Overall Study
Arm/Group | Depacon IV and Depakote
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Depacon IV and Depakote
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Time Required to Achieve a Greater Than or Equal to 50% Reduction in Frequency or Severity of Individual Cluster Attacks Compared to Subject-reported Baseline.
Description: Severity: measured on an 11 point scale, where 0 = no pain and 10= excruciating pain. Outcome is time to 50% reduction in severity (or frequency) compared to baseline (prior to treatment).Frequency: Number of attacks per day.The Time to significant response was measured 2 ways: significant initial response and significant maintained response. For initial response, the time to significant response was: Mean of 2.1(1.5) days for severity and 1.9 (1.6) days for frequency. The time to significant response maintained was 29.7 (13.8) for severity and 29.0 (14.3) for frequency.
Time Frame: baseline (day 0) through 47 days after first infusion
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Depacon IV and Depakote
Number analyzed (Participants) | 15
days | 29.7 (13.8)

2. Secondary Outcome: Change in Frequency of Attacks Per 24 Hour Period, Duration of Individual Attacks (in Minutes), or Severity of Attacks Compared to the Subject-reported Baseline Values.
Time Frame: Compare Baseline through 47 days
Reporting Status: Not Posted
Measure: Number (Standard Deviation); unit: days

3. Secondary Outcome: Use of Acute and Rescue Medications During Loading (2 Days) and Maintenance Phases as Compared to Subject-reported Baseline. This Will be Calculated Using the Total Number of Doses of Acute Medications Per 24-hour Period Calendar Days.
Time Frame: Baseline compared to maintenance (up to 47 days)
Reporting Status: Not Posted
Measure: Number (Standard Deviation); unit: number doses

ADVERSE EVENTS:
Arm/Group | Depacon IV and Depakote
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 7/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Depacon IV and Depakote (N=15)
cool sensation (Metabolism and nutrition disorders) | 2 — Cool sensation during infusion
Tiredness (Nervous system disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Taste perversion (Nervous system disorders) | 1
Warm sensation (Nervous system disorders) | 1
Lightheadedness (Nervous system disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes